CLINICAL TRIAL: NCT03190278
Title: Phase I, Open Label Dose Escalation and Dose-Expansion Study to Evaluate the Safety, Expansion, Persistence, and Clinical Activity of UCART123 (Allogeneic Engineered T-cells Expressing Anti-CD123 Chimeric Antigen Receptor), Administered in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Study Evaluating Safety and Efficacy of UCART123v1.2 in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Acronym: AMELI-01
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cellectis S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCART123_01
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Relapsed/Refractory Acute Myeloid Leukemia; Chimeric Antigen Receptor T-Cell (CAR-T) therapy; Allogeneic; Transcription Activator-Like Effector Nuclease (TALEN)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): UCART123v1.2 tested at several dose levels with different lymphodepletion regimens to establish Maximum Tolerated Dose (MTD) and identify Recommended Phase 2 Dose (RP2D)
  Dose Expansion: UCART123v1.2 administered at the RP2D determined from the dose escalation phase
  Interventions: Biological: UCART123v1.2

INTERVENTIONS:
Biological: UCART123v1.2 — Allogeneic engineered T-cells expressing anti-CD123 Chimeric Antigen Receptor Biological/vaccine: CLLS52 A monoclonal antibody that recognizes the CD52 antigen Other Names: Alemtuzumab

SUMMARY:
Phase I, open-label, dose-escalation and dose-expansion study evaluating the safety and efficacy of Universal Chimeric Antigen Receptor T-cell (UCART) targeting the Cluster of Differentiation 123 (CD123) in patients with relapsed/refractory acute myeloid leukemia (AML). The purpose of this study is to evaluate the safety and clinical activity of Universal Chimeric Antigen Receptor T-cells targeting CD123 (UCART123v1.2) and determine the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D).

ELIGIBILITY:
Main Inclusion Criteria:

* Patients with relapsed or primary refractory AML (as defined in World Health Organization [WHO] criteria) with ≥5% bone marrow blasts
* Patients with CD123+ blast cells (verified by flow cytometry)
* Eastern Cooperative Oncology Group Performance Status (ECOG-PS) of ≤1
* Adequate organ function, including bone marrow, renal, hepatic, pulmonary, and cardiac function based on the last assessment performed within screening period
* (Dose-escalation) Identified donor and transplant strategy prior to lymphodepletion (LD)
* Other criteria may apply

Main Exclusion Criteria:

* Patients with acute promyelocytic leukemia (APL) or central nervous system (CNS) Leukemia
* Previous investigation gene or cell therapy (including CAR)
* > 1 prior allogeneic stem cell transplantations (SCTs)
* Prior treatment with rituximab or other anti-cluster of differentiation 20 (anti-CD20) therapy within 3 months
* Any known active or uncontrolled infection
* Other criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AE)/serious adverse events (SAE)/Dose Limiting Toxicities (DLT) [Safety and Tolerability] | 24 Months
  Safety of UCART123v1.2 - Incidence, nature, and severity of AE and SAEs throughout the study
Dose escalation and expansion part: Occurrence of DLTs | Up to Day 28 post last UCART123v1.2 infusion

SECONDARY OUTCOMES:
Investigators assessed overall response rate according to the European Leukemia Net (ELN) Response Criteria | At Day 28, Day 56, Day 84, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 21 and Month 24
Duration of Response | From the date of the initial response to the date of disease progression or death from any cause, whichever occurs first, assessed up to Month 24
Progression Free Survival | From the first day of study treatment to the date of disease progression or death from any cause, whichever occurs first, assessed up to Month 24
Overall Survival | From the first day of study treatment to the date of death from any cause, assessed up to Month 24
Pharmacokinetic (PK) Analysis: Standard PK Analysis will be completed to obtain Maximum plasma concentration (Cmax) | alemtuzumab levels will be determined pre- and post-dose alemtuzumab and up to 48 hours after the last dose
Pharmacokinetic Analysis: Standard PK Analysis will be completed to obtain time to reach Cmax (Tmax) | alemtuzumab levels will be determined pre- and post-dose alemtuzumab and up to 48 hours after the last dose
Pharmacokinetic Analysis: Standard PK Analysis will be completed to obtain total area under curve from zero to infinity (AUC-infinity) | alemtuzumab levels will be determined pre- and post-dose alemtuzumab and up to 48 hours after the last dose
Pharmacokinetic Analysis: Standard PK Analysis will be completed to obtain Terminal Rate | alemtuzumab levels will be determined pre- and post-dose alemtuzumab and up to 48 hours after the last dose
Pharmacokinetic Analysis: Standard PK Analysis will be completed to obtain Terminal Half-life | alemtuzumab levels will be determined pre- and post-dose alemtuzumab and up to 48 hours after the last dose
Pharmacokinetic Analysis: Standard PK Analysis will be completed to obtain Clearance | alemtuzumab levels will be determined pre- and post-dose alemtuzumab and up to 48 hours after the last dose
Pharmacokinetic Analysis: Standard PK Analysis will be completed to obtain Volume of Distribution | alemtuzumab levels will be determined pre- and post-dose alemtuzumab and up to 48 hours after the last dose
Pharmacodynamic Analysis: Pharmacodynamics Monitoring of the incidence of anti-cluster of differentiation 52 (anti-CD52; alemtuzumab) antibodies (ADA) in serum Pre-alemtuzumab administration and through Day 84 | From screening through Day 84
Pharmacodynamic Analysis: Pharmacodynamics Quantitation of T cells in peripheral blood | From screening through Day 84
Pharmacodynamic Analysis: Pharmacodynamics Quantitation of B cells in peripheral blood | From screening through Day 84
Pharmacodynamic Analysis: Pharmacodynamics Quantitation of natural killer (NK) cells in peripheral blood | From screening through Day 84
Pharmacodynamic Analysis: Pharmacodynamics Quantitation of total lymphocytes in peripheral blood | From screening through Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Gail Roboz, Dr, Principal Investigator — Weill Medical College of Cornell University
Locations (8):
- United States (8):
  - University of California, San Francisco (UCSF) - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of Pennsylvania - Abramson Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No